CLINICAL TRIAL: NCT04682028
Title: Construction and Evaluation a Network Platform of Continuous Care for Ostomy Patients
Brief Title: Construction and Evaluation of a Stoma Patient Continuous Care Network
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XJTU1AF2020LSK-228
Record Dates: First submitted 2020-12-20; First posted 2020-12-23 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-08

CONDITIONS: Surgical Stomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Other): Nurses provide web-based continuous care to patients.
  Interventions: Other: professional care
- contral group (Other): Nurses provide the routine care to patients.
  Interventions: Other: coventional care

INTERVENTIONS:
Other: professional care — The trained nurses provide professional care for the patients.
  Arms: experiment group
Other: coventional care — nurses provide coventional care for the patients.
  Arms: contral group

SUMMARY:
Construct a professional network platformof continuous care for patients with enterostomy and evaluate its availability， Eventually, patients with enterostomy will have access to care outside the hospital.

DETAILED DESCRIPTION:
The project to establish a professional care network for stomas patient will be conducted at first Affiliated Hospital Xi'an Jiaotong University.This network platform that patients can enjoy to make an appointment, video interrogation, the inspection booking, self management, health education, and other health and extension services;nursing staff can undertake colostomy online learning and assessment of the relevant knowledge and skills;professional colostomy care is published to provide remote guidance.the efficacy of the network was evaluated by investigating complications rate,and their self-care ability,quality of life, and medical expenses,and patients'satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patients aged≥18 years old;
* patients undergoing enterostomy;
* patients possess a smart phone and know how to use it;
* patients volunteer to participate in the survey.

Exclusion Criteria:

* patients have a history of mental disorders;
* cancer has metastasized to other organs, or there are other serious physical diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
stomy Quality of Life,Stoma-QOL | up to 9 months
  The scale includes 20 items with a score ranging from 20 to 80points.The higher the score,the better the quality of life.

SECONDARY OUTCOMES:
Enterostomy Patients Self-management Questionnaire | up to 9 months
  The scale includes 5 dimensions,30items;The higher the score,the better the Self-management.
Stoma and surrounding complications | up to 9 months
  Stoma complications include infection around the stoma,skin and mocous membrane separation, hemorrhage etal.

CONTACTS AND LOCATIONS:
Overall Officials: Xiulin Wen, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- first Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No